CLINICAL TRIAL: NCT04082585
Title: Total Health Improvement Program Research Project (A Community Lifestyle Medicine Course and Ability to Improve Health in All Classes of Socioeconomic Status)
Brief Title: Total Health Improvement Program Research Project
Status: Completed | Type: Observational
Sponsor: Pacific Northwest University of Health Sciences (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Better Living Center (Unknown)
Responsible Party: Principal Investigator, Heidi Beery, Principal Investigator, Pacific Northwest University of Health Sciences
Other Study IDs: 2019-019
Record Dates: First submitted 2019-08-28; First posted 2019-09-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Chronic Disease; Cardiovascular Diseases; Hypertension; Diabetes; Pre-diabetes; Obesity
MeSH Terms: conditions — Chronic Disease; Cardiovascular Diseases; Hypertension; Diabetes Mellitus; Glucose Intolerance; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Total Health Improvement Program — The Total Health Improvement program is a 13 week community based nutrition program designed to assist participants in improving their physical and emotional well being. The program focuses on a plant based diet and increased physical activity.

SUMMARY:
The purpose of this study is to assess the effectiveness a 13-week community based nutrition education program to assist participants program in improving in physical and emotional well being and to assess if there are differences in outcomes based on a participant's socioeconomic status.

DETAILED DESCRIPTION:
Little is known about effective strategies to reduce inequalities in non-communicable diseases (NCDs) and their underlying behaviors. McGill et al did a systematic review of the socioeconomic inequalities in promoting healthy eating. They found that upstream interventions with policy changes on price (fiscal measures such as taxes, subsidies, or economic incentives) reduced socioeconomic inequalities compared to downstream interventions such as cooking lessons, tailored nutritional education/counseling or nutrition education in the school curriculum appear likely to widen inequalities.

Douglas County's average income is $44,023 (compared to the median annual income of $60,336 across the entire United States) and the 5th poorest county in the state. 17% of the population is in poverty, higher than the national average of 13.4%.

The Complete Health Improvement Program (CHIP) is a premier lifestyle intervention that has been offered for more than 25 years and has been shown in over 25 peer-reviewed publications to benefit chronic disease. The Complete Health Improvement Program (CHIP) is a premier lifestyle intervention that has been offered for more than 25 years and has been shown in over 25 peer-reviewed publications to benefit chronic disease. CHIP was initially offered in Douglas County 5 years ago and found to benefit participants but there were concerns that it was widening inequalities due to the cost of the class. A similar program named Total Health Improvement Program (THIP) was designed and offered to the community for free through the partnership of a non-profit organization called UC-VEG.

The purpose of this study is to determine the effectiveness of the 13-week community-based nutrition education THIP program to assist participants with the adoption of a plant-based diet, increase physical activity and increase positive psychology. Research has shown plant-based diets to be safe and effective for weight management or reduction, cholesterol management, hypertension and diabetes management, and overall health and longevity. The primary objectives are to assess the effectiveness of the program in improving physical and emotional well-being and to assess if there are differences in outcomes based on a participant's socioeconomic status.

ELIGIBILITY:
Inclusion Criteria:

* Speak English
* 18 years of age or older
* Prepared to engage in the Total health Improvement Program (THIP) weekly educational classes (13 weeks)
* Willing to participate in the pre and post questionnaire
* Able to participate in the lab work at weeks 2 and 12
* Have at least one chronic disease including cardiovascular disease, hyperlipidemia, hypertension, obesity (BMI >30), diabetes, or pre-diabetes (A1C>5.7%)
* Able to provide their own meals (whole foods diet)
* Has not attended the THIP program in the last year

Exclusion Criteria:

* Non English Speakers
* Less than 18 years of age
* Unwilling to engage in the Total health Improvement Program (THIP) weekly educational classes (13 weeks)
* Unwilling to participate in the pre and post questionnaire
* Not able to participate in the lab work at weeks 2 and 12
* Do not have at least one chronic disease including cardiovascular disease, hypertension, diabetes or pre-diabetes (A1C>5.7%)
* Unable to provide their own meals (whole foods diet)
* Has attended the THIP program in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have at least one chronic disease and may or maynot be economically or educationally disadvantaged.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline - Global Health Score | 12 weeks
  Change in global health score as measured by the validated SF-20 survey. The survey is scored for limitations in physical and role functioning (a higher score value indicates better functioning, for mental health (a higher score value indicates better health) and for pain (a higher score value indicates more pain).
Correlation of Global Health Scores to Social Determinants of Health | 12 weeks
  The primary analysis will be to determine if changes in SF-20 score are correlated with scores from the PCS3 Socioeconomic Survey to determine the relationship, if any, between socioeconomic status and changes in global health.

SECONDARY OUTCOMES:
Change from Baseline - Weight | 12 Weeks
  The participants will be weighed at week 2 (baseline) and week 12. The data will be analyzed to determine effectiveness of the Total Health Improvement Program.
Change from Baseline - Abdominal Circumference | 12 Weeks
  The participants will have there abdominal circumference measured at week 2 (baseline) and week 12. The data will be analyzed to determine effectiveness of the Total Health Improvement Program.
Change from Baseline - HbA1C | 12 Weeks
  The participants will have blood draws at week 2 (baseline) and week 12 and results will be compared to determine effectiveness of the Total Health Improvement Program. .
Change from Baseline - Total Cholesterol | 12 Weeks
  The participants will have blood draws at week 2 (baseline) and week 12 and results will be compared to determine effectiveness of the Total Health Improvement Program. .
Change from Baseline - Triglycerides | 12 Weeks
  The participants will have blood draws at week 2 (baseline) and week 12 and results will be compared to determine effectiveness of the Total Health Improvement Program. .
Change from Baseline - LDL Cholesterol | 12 Weeks
  The participants will have blood draws at week 2 (baseline) and week 12 and results will be compared to determine effectiveness of the Total Health Improvement Program. .
Change from Baseline - HDL Cholesterol Ratio | 12 Weeks
  The participants will have blood draws at week 2 (baseline) and week 12 and results will be compared to determine effectiveness of the Total Health Improvement Program. .

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Beery, MD, Principal Investigator — Pacific Northwest University of Health Science
Locations (1):
- Better Living Center, Roseburg, Oregon, United States

IPD SHARING:
Plan to Share IPD: No